CLINICAL TRIAL: NCT07316621
Title: Prospective Risk Evaluation and Detection of Crohn's Disease in First-degree Relatives
Acronym: PREDICT-CD
Status: Not yet recruiting | Type: Observational
Sponsor: GLSMED Learning Health S.A. (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT-CD
Record Dates: First submitted 2025-12-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First-degree relatives

SUMMARY:
The PREDICT-CD study aims to validate a risk score for the development of Crohn's disease, based on serological biomarkers and lifestyle-related factors. Given that having a family member with the disease is the strongest known risk factor, the target population will consist of first-degree relatives (aged 16 to 35) of individuals diagnosed with Crohn's disease.

This study will be conducted within Work Package 3 (WP3) of the INTERCEPT project, a consortium funded by the Innovative Health Initiative (IHI). The research will take place across 28 centres in seven countries: Portugal, Spain, France, Italy, the Netherlands, Sweden, and Poland.

To achieve the study objectives, individuals with Crohn's disease (referred to as patients) will be invited to participate and to engage their eligible first-degree relatives. At the baseline visit, the patient's physician will complete a clinical questionnaire covering disease history, treatments, and previous interventions.

At the same time, first-degree relatives (parents, siblings, or children) will donate a blood sample for serum isolation and, optionally, a whole blood and stool sample. They will also complete a questionnaire regarding their health status, habits, and preferences. Follow-up questionnaires will be administered every six months to monitor the onset of symptoms or behavioural changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, between 16 and 35 years old
* FDR (parent, full-siblings or offspring) from a patient with an established diagnosis of CD
* Participants able to understand the information provided to them and to give written informed assent or consent for the study.

Exclusion Criteria:

* Prior diagnosis of IBD
* Any legal or medical condition that limits the information and participation in the study
* Inability to verify CD diagnosis in the proband
* Participants unwilling or unable to provide informed written consent
* Participants unwilling or unable to donate blood for serum

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The first-degree relative without a previous diagnosis of Inflammatory Bowel Disease
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the performance of a risk model for at-risk population for CD | through study development, an average of 1-3 year
  The model will integrate measures of predefined serum biomarkers of at-risk population (first degree relatives of CD patients) with clinical and lifestyle factors. The performance can than be assessed by the risk prediction of participants which are then diagnosed with CD.

SECONDARY OUTCOMES:
Prevalence of risk factors in FDRs developing IBD | throughout the study, in average 1-3 years
  Evaluation of early life risk factors, dietary and nutritional patterns, fatigue, stress, and physical exercise levels, smoking history and exposure to smoking, medical and surgical history, and medication history in FDRs developing IBD during the study through semestral questionnaires

IPD SHARING:
Plan to Share IPD: No